CLINICAL TRIAL: NCT00872833
Title: Assessment of Pain in Transfusion Dependent Patients With Thalassemia During Transfusion Cycles
Brief Title: Assessment of Pain in People With Thalassemia Who Are Treated With Regular Blood Transfusions
Status: Completed | Type: Observational
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 640; U01HL065238 (NIH)
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Results first posted 2014-08-27 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2012-04

CONDITIONS: Thalassemia
Keywords: Transfusion-Dependant Thalassemia; Pain; Mild Pain
MeSH Terms: conditions — Thalassemia; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- age 18-29: People age groups 18-29 with transfusion-dependent thalassemia who have reported at least mild degrees of pain during the main Assessment of Pain study.
- age 30+: People age groups 30+ years with transfusion-dependent thalassemia who have reported at least mild degrees of pain during the main Assessment of Pain study.

SUMMARY:
Thalassemia is an inherited blood disorder that can result in mild to severe anemia. Regular blood transfusions, which refresh the healthy red blood cell supply, are one treatment for thalassemia. People with thalassemia often experience pain, but the exact source of pain remains unknown. This study will examine how pain varies during the blood transfusion cycle in people with thalassemia who are treated with regular blood transfusions.

DETAILED DESCRIPTION:
Thalassemia is an inherited blood disorder in which the body makes an abnormal form of hemoglobin-the protein in red blood cells that carries oxygen. People with thalassemia often experience fatigue, shortness of breath, and pain. There have been no previous research studies that have fully examined pain levels in people with thalassemia, and as a result, the sources of pain remain unknown. This study is a substudy of the Assessment of Pain study, which is a Thalassemia Clinical Research Network (TCRN) study that is examining the prevalence and severity of pain in people with transfusion-dependent thalassemia and non-transfusion-dependant thalassemia. This study will enroll a subset of participants from the Assessment of Pain study who have transfusion-dependant thalassemia. The purpose of this study is to examine whether pain varies during the blood transfusion cycle and whether the length of the transfusion cycle affects pain levels in people with transfusion-dependent thalassemia.

Participants will complete daily questionnaires through an automated telephone system to assess pain levels during three blood transfusion cycles. Each transfusion cycle will last between 2 to 4 weeks, depending on the individual needs of the participant, and the cycles will be separated by at least 3 months but no more than 4 months. Prior to each transfusion cycle, study researchers will review participants' medical records for certain blood level measurements.

ELIGIBILITY:
Inclusion Criteria:

* Participating in the Thalassemia Clinical Research Network Assessment of Pain study
* Has a transfusion dependence of at least eight transfusions per year
* Diagnosis of beta thalassemia or E-beta-thalassemia
* Experiences at least "mild" pain in the 1 month before study entry, as measured by the response to the Brief Pain Inventory (BPI) question #6 from the Assessment of Pain study

Exclusion Criteria:

* Unwillingness or inability to complete the Brief Pain Inventory Short Form (BPI-SF) on a daily basis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with transfusion-dependent thalassemia who receive care at sites funded by the Thalassemia Clinical Research Network and their satellites.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2009-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dru Foote, NP, Principal Investigator — Children's Hospital and Research Institute Oakland; Jeanne Boudreaux, MD, Study Chair — Children's Healthcare of Atlanta; Thomas Coates, MD, Study Chair — Children's Hospital Los Angeles; Elliott Vichinsky, MD, Study Chair — UCSF Benioff Children's Hospital Oakland; Michael Jeng, MD, Study Chair — Stanford University; Janet Kwiatkowski, MD, Study Chair — Children's Hospital of Philadelphia; Nancy Olivieri, MD, Study Chair — University Health Network - Toronto General Hospital; Patricia J. Giardina, MD, Study Chair — Weill Medical College of Cornell; Brigitta Mueller, MD, Study Chair — Baylor College of Medicine; Alexis A. Thompson, MD, MPH, Study Chair — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (9):
- United States (8):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital Research Center Oakland, Oakland, California
  - Stanford University - School of Medicine, Stanford, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Weill Medical College of Cornell, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
- University Health Network - Toronto General Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Younger Cohort: People age groups 18-29 with transfusion-dependent thalassemia who have reported at least mild degrees of pain during the main Assessment of Pain study.
- Older Cohort: People age groups 30+ years with transfusion-dependent thalassemia who have reported at least mild degrees of pain during the main Assessment of Pain study.
Period: Overall Study
Arm/Group | Younger Cohort | Older Cohort
Started | 15 | 17
Completed | 15 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: Both cohorts combined
Arm/Group | Overall
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Report of Pain by Age Group
Description: Subjects reported whether or not they had pain (yes/no) during each transfusion cycle (data on up to 3 transfusion cycles were collected for each subject). The percent of subject-cycles with pain was calculated for the quartiles of the transfusion cycle.
Time Frame: measured daily over the 3 transfusion cycles
Measure: Number; unit: percentage of participant-cycles
Units Other Than Participants: Participant-cycles
Arm/Group | Younger Cohort | Older Cohort
Number analyzed (Participants) | 15 | 17
Number analyzed (Participant-cycles) | 40 | 43
percentage of participant-cycles
  Start of cycle | 23 | 61
  25% through cycle | 18 | 51
  50% through cycle | 15 | 47
  75% through cycle | 20 | 54
  End of cycle | 18 | 56
Statistical Analysis 1: Comparison: Younger Cohort vs Older Cohort; Test type: Superiority or Other; p < .001, Chi-squared

2. Secondary Outcome: Report of Pain by Length of the Transfusion Cycle
Description: as for outcome 1
Time Frame: measured daily over the 3 transfusion cycles
Population: Unit of analysis was participant-cycle. Data were collected over (at most) three transfusion cycles for each subject. Transfusion cycle lengths varied, and subjects may be represented in more than one arm/group.
Measure: Number; unit: percentage of participant-cycles
Units Other Than Participants: Participant-cycles
Groups:
- <= 14 Days: Subjects with transfusion cycles of 14 days or less
- 15 - 21 Days: Subjects with transfusion cycles between 15 and 21 days
- 22 - 28 Days: Subjects with transfusion cycles between 22 and 28 days
- > 28 Days: Subjects with transfusion cycles greater than 28 days
Arm/Group | <= 14 Days | 15 - 21 Days | 22 - 28 Days | > 28 Days
Number analyzed (Participants) | 5 | 12 | 17 | 13
Number analyzed (Participant-cycles) | 10 | 25 | 26 | 22
percentage of participant-cycles
  Start of cycle | 50 | 40 | 42 | 41
  25% through cycle | 50 | 48 | 35 | 14
  50% through cycle | 50 | 48 | 23 | 14
  75% through cycle | 60 | 52 | 31 | 18
  End of cycle | 50 | 44 | 31 | 32
Statistical Analysis 1: Comparison: <= 14 Days vs 15 - 21 Days vs 22 - 28 Days vs > 28 Days; Test type: Superiority or Other; p = 0.028, Chi-squared

ADVERSE EVENTS:
Description: Adverse event data were not collected for this observational study
Groups:
- Adverse Events Were Not Collected: Adverse events were not collected as part of this observational study.
Arm/Group | Adverse Events Were Not Collected
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No